CLINICAL TRIAL: NCT02061280
Title: Use of Mobile Devices and the Internet to Streamline an Asthma Clinical Trial
Acronym: MICT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 332965; R01HL114899 (NIH)
Record Dates: First submitted 2014-01-31; First posted 2014-02-12 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Asthma
Keywords: Asthma; Clinical Trial Design; Electronic Data Entry; Mobile Devices; Home Spirometry
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination; Dry Powder Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MICT Trial Design (Experimental): Participants randomized to MICT will complete study procedures using an iPad for data entry and FaceTime visits rather than coming into the study site for onsite visits. Participants will perform spirometry at home using a handheld spirometer, EasyOne Plus.
  Randomized to one of 3 study treatments:
  fluticasone/salmeterol 250/50 Dry Powder Inhaler one inhalation twice daily, or fluticasone/salmeterol 100/50 Dry Powder Inhaler one inhalation twice daily, or fluticasone 100mcg Dry Powder Inhaler one inhalation twice daily
  Interventions: Drug: fluticasone/salmeterol 250/50 Dry Powder Inhaler; Drug: fluticasone/salmeterol 100/50 Dry Powder Inhaler; Drug: fluticasone 100mcg Dry Powder Inhaler
- LASST Trial Design (Active Comparator): Participants randomized to LASST will complete study procedures in the traditional format in which all study visits are conducted at the study site, all questionnaires are completed by pen/paper, and all spirometry is performed at the clinic site.
  Randomized to one of 3 study treatments:
  fluticasone/salmeterol 250/50 Dry Powder Inhaler one inhalation twice daily, or fluticasone/salmeterol 100/50 Dry Powder Inhaler one inhalation twice daily, or fluticasone 100mcg Dry Powder Inhaler one inhalation twice daily.
  Interventions: Drug: fluticasone/salmeterol 250/50 Dry Powder Inhaler; Drug: fluticasone/salmeterol 100/50 Dry Powder Inhaler; Drug: fluticasone 100mcg Dry Powder Inhaler

INTERVENTIONS:
Drug: fluticasone/salmeterol 250/50 Dry Powder Inhaler — Participants will receive Advair Diskus 250/50 Dry Powder Inhaler, administered twice daily for 12 weeks after randomization
  Other Names: Advair Diskus
Drug: fluticasone/salmeterol 100/50 Dry Powder Inhaler — Participants will receive Advair Diskus 100/50 Dry Powder Inhaler administered twice daily for 12 weeks after randomization
  Other Names: Advair Diskus
Drug: fluticasone 100mcg Dry Powder Inhaler — Participants will receive Flovent Diskus 100mcg Dry Powder Inhaler administered twice daily for 12 weeks after randomization
  Other Names: Flovent Diskus

SUMMARY:
Asthma is an inflammatory disease that imposes a significant burden affecting an estimated 300 million persons and 20% of all children worldwide. It is one of the most common chronic diseases of childhood and is a leading cause of school absenteeism. There continues to be a great need for clinical trials in asthma but traditional clinical trials are expensive and reasons cited by patients for non-participation are extra inconvenience and logistical barriers. Study designs which are patient centered and reduce trial costs are needed. The long-range goal of this application is to transform the paradigm of clinical research into a more efficient and cost-effective enterprise by capitalizing upon current widely used mobile electronic means of communication and information transfer.

This innovative project is a streamlined clinical trial that will run concurrently with a nearly identical traditional clinical trial, "Long-acting Beta Agonist Step Down Study" (LASST) which will allow for direct comparison of processes and outcomes between the streamlined and traditional approach. Children 12 to 17 years old with asthma will be randomized to participate in this project (streamlined trial) or LASST (traditional trial). In this proposal we will: measure comprehension of study information using an original questionnaire, Research Participant Assessment (developed at Nemours), following a parental permission/assent process delivered over the internet in a dynamic interactive multi-media format (Specific Aim 1); measure the efficiency of participant driven data entry from home into a Research Electronic Data Capture (REDCap) online database using the iPad, and quality of spirometry with the EasyOne Plus handheld meter with remote coaching using the iPad (Specific Aim 2); test whether the streamlined approach has a "trial effect" by comparing the differences in Asthma Control Test (ACT) scores following 12 weeks of study drug treatment in children randomized to this project compared to LASST. We will collect effort reporting data to compare personnel costs between the trials. If this streamlined project lacks a "trial effect" and reduces costs compared to LASST, the methodologies would be generalizable to studies which include adults and other diseases.

DETAILED DESCRIPTION:
Introduction Phase III / IV clinical trials are expensive and time consuming and often suffer from poor enrollment and retention rates. Pediatric trials are particularly difficult because scheduling around the parent, participant and potentially other sibling schedules can be burdensome. We are evaluating using the internet and mobile devices to conduct the consent process and study visits in a streamlined pediatric asthma trial. Our hypothesis is that these study processes will be noninferior and will be less expensive compared to a traditional pediatric asthma trial.

Materials/Methods Parents and participants, aged 12 through 17 years, complete the informed consent process by viewing a multi-media website containing a consent video and study material in the streamlined trial. Participants are provided an iPad with WiFi (wireless internet) and EasyOne spirometer for use during FaceTime visits and online twice daily symptom reporting during an 8-week run-in followed by 12-week study period. Outcomes are compared with participants completing a similarly designed traditional trial comparing the same treatments within the same pediatric health-system. After 8 weeks of open-label Advair 250/50 twice daily, participants in both trial types are randomized to Advair 250/50, Flovent 250, or Advair 100/50 given 1 inhalation twice daily. Study staff track time spent to determine study costs.

Results Participants have been enrolled in the streamlined and traditional trials and recruitment is ongoing.

Conclusions This project will provide important information on both clinical and economic outcomes for a novel method of conducting clinical trials. The results will be broadly applicable to trials of other diseases.

ELIGIBILITY:
Main Trial

Inclusion Criteria:

* Age 12-17 years
* Physician diagnosed asthma (without any other co-morbid pulmonary disease) that is well-controlled on medium dose inhaled corticosteroid and long-acting β2-agonist given twice daily [Advair Diskus (fluticasone propionate/salmeterol) 250/50mcg; Advair HFA (hydrofluoroalkane) (fluticasone propionate/salmeterol hydrofluoroalkane) 115/21mcg; Symbicort (budesonide/formoterol) 160/4.5mcg; Dulera (mometasone/formoterol) 100/4.5mcg] based on an ACT score > 20, and the absence of unscheduled visits or use of rescue prednisone for 4 weeks prior to enrollment
* Pre-bronchodilator forced expiratory volume in the first second > 70% predicted
* < 10 pack/year history of tobacco use and abstinence for at least 1 year

Exclusion Criteria:

* Chronic oral steroid therapy
* Hospitalization or urgent care visit within 4 weeks of the screening visit
* Near fatal asthma within 2 years of enrollment or high risk of near fatal or fatal asthma 125-127
* Women who are pregnant or lactating

Parallel MICT and Parallel LASST

Inclusion Criteria:

* Age 12-17 years
* Physician diagnosed asthma (without any other co-morbid pulmonary disease) that is well-controlled on medium dose inhaled corticosteroid and long-acting β2-agonist given twice daily [Advair Diskus (fluticasone propionate/salmeterol) 250/50mcg; Advair HFA (hydrofluoroalkane) (fluticasone propionate/salmeterol hydrofluoroalkane) 115/21mcg; Symbicort (budesonide/formoterol) 160/4.5mcg; Dulera (mometasone/formoterol) 100/4.5mcg] based on an ACT score > 20, and the absence of unscheduled visits or use of rescue prednisone for 4 weeks prior to enrollment
* < 10 pack/year history of tobacco use and abstinence for at least 1 year

Exclusion Criteria:

* Chronic oral steroid therapy
* Hospitalization or urgent care visit within 4 weeks of the screening visit
* Near fatal asthma within 2 years of enrollment or high risk of near fatal or fatal asthma 125-127
* Women who are pregnant or lactating

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2013-10; Primary Completion 2017-02-17 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Blake, PharmD, Principal Investigator — Nemours Children's Clinic Jacksonville FL
Locations (5):
- United States (5):
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Specialty Care, Pensacola, Florida
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Deidentified datasets, study forms, study protocol, study manual of procedures will be deposited into BioLINCC.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be deposited in BioLINCC after the primary manuscript is published which is expected to be by January 2019.
Access Criteria: Requests for access to data will be in accordance with any requirements set forth by BioLINCC.

REFERENCES:
- [Background] Blake K, Holbrook JT, Antal H, Shade D, Bunnell HT, McCahan SM, Wise RA, Pennington C, Garfinkel P, Wysocki T. Use of mobile devices and the internet for multimedia informed consent delivery and data entry in a pediatric asthma trial: Study design and rationale. Contemp Clin Trials. 2015 May;42:105-18. doi: 10.1016/j.cct.2015.03.012. Epub 2015 Apr 3. PMID 25847579
- [Background] Antal H, Bunnell HT, McCahan SM, Pennington C, Wysocki T, Blake KV. A cognitive approach for design of a multimedia informed consent video and website in pediatric research. J Biomed Inform. 2017 Feb;66:248-258. doi: 10.1016/j.jbi.2017.01.011. Epub 2017 Jan 19. PMID 28109951
- [Derived] Blake KV, Antal H, Bunnell HT, He J, Henderson R, Holbrook JT, McCahan SM, Pennington C, Rogers L, Shade D, Sugar EA, Taylor A, Wise RA, Wysocki T. Comprehension by Caregivers and Adolescents of Clinical Trial Information Delivered via Multimedia Video Versus Conventional Practice: Nonrandomized Controlled Trial. JMIR Pediatr Parent. 2023 Jun 22;6:e44252. doi: 10.2196/44252. PMID 37347518

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MICT Trial Design | LASST Trial Design
Started (Individuals who signed informed consent form.) | 71 | 37
Randomized to Treatment (Individuals randomized to drug treatment at Visit 3.) | 54 | 25
Completed | 53 | 25
Not Completed | 18 | 12
Not completed — Protocol Violation | 12 | 8
Not completed — moved out of state | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Population: 54 participants in the MICT trial arm were randomized to drug treatment at Visit 3, 53 participants completed the Visit 6 (final) Consent Assessment Interview.
  25 participants in the LASST trial were randomized to drug treatment at Visit 3; 25 participants completed the Visit 6 (final) Consent Assessment Interview.
Groups:
- Total: Total of all reporting groups
Arm/Group | MICT Trial Design | LASST Trial Design | Total
Number analyzed (Participants) | 54 | 25 | 79
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [13 to 15] | 15 [13 to 16] | 14 [13 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 12 | 34
  Male | 32 | 13 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 2 | 51
  Not Hispanic or Latino | 5 | 23 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 10 | 26
  White | 30 | 15 | 45
  More than one race | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 25 | 79
Unscheduled Health Care Visit in Past 12 Months [Count of Participants; unit: Participants] | 23 | 9 | 32

OUTCOME MEASURES:

1. Primary Outcome: Adolescent Research Participant Assessment Score at Screening (Visit 1, Week -8)
Description: The Research Participant Assessment Score (RPA Comprehension) was a 17-item questionnaire designed to assess comprehension of study information at screening (Visit 1, week -8) between MICT and LASST trial designs. The same 17-item questionnaire was administered to the adolescent participant and to the caregiver participant. The items were scored as 1=incorrect, 2=partially correct, 3=correct (minimum possible score=17 and maximum possible score=51). Scores were assigned by two trained coders who independently listed to audio recordings of the RPA Comprehension questionnaire administration. Scores from the two coders were averaged for a final score. Higher scores indicate better comprehension. Mean (95% Confidence Interval) are the outcome measure reported.
Time Frame: Screening (Visit 1, week -8)
Population: One participant in the MICT trial arm who was randomized to treatment at Visit 3 did not complete the study through Visit 6.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- MICT Trial Design: Participants randomized to MICT will complete study procedures using an iPad for data entry and FaceTime visits rather than coming into the study site for onsite visits. Participants will perform spirometry at home using a handheld spirometer, EasyOne Plus.
  Randomized to one of 3 study treatments:
  fluticasone/salmeterol 250/50 Dry Powder Inhaler one inhalation twice daily fluticasone/salmeterol 100/50 Dry Powder Inhaler one inhalation twice daily fluticasone 100mcg Dry Powder Inhaler one inhalation twice daily
- LASST Trial Design: Participants randomized to LASST will complete study procedures in the traditional format in which all study visits are conducted at the study site, all questionnaires are completed by pen/paper, and all spirometry is performed at the clinic site.
  Randomized to one of 3 study treatments:
  fluticasone/salmeterol 250/50 Dry Powder Inhaler one inhalation twice daily fluticasone/salmeterol 100/50 Dry Powder Inhaler one inhalation twice daily fluticasone 100mcg Dry Powder Inhaler one inhalation twice daily
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 53 | 25
Scores on a scale | 41.08 [39.48 to 42.69] | 42.26 [39.9 to 44.62]

2. Primary Outcome: Caregiver Research Participant Assessment Score at Screening (Visit 1, Week -8)
Description: as for outcome 1
Time Frame: Screening (Visit 1, week -8)
Population: One participant in the MICT trial arm who was randomized to treatment at Visit 3 did not complete the study through Visit 6. Thus, the caregiver did not complete the Research Participant Assessment at Visit 6.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- MICT Trial Design: MICT Trial:
  Participants randomized to MICT will complete study procedures using an iPad for data entry and FaceTime visits rather than coming into the study site for onsite visits. Participants will perform spirometry at home using a handheld spirometer, EasyOne Plus.
  Randomized to one of 3 study treatments:
  fluticasone/salmeterol 250/50 Dry Powder Inhaler one inhalation twice daily fluticasone/salmeterol 100/50 Dry Powder Inhaler one inhalation twice daily fluticasone 100mcg Dry Powder Inhaler one inhalation twice daily
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 53 | 25
Scores on a scale | 43.2 [41.96 to 44.45] | 42.9 [41.06 to 44.74]

3. Secondary Outcome: Adolescent Research Participant Assessment Score at Study End (Visit 6, Week 12)
Description: The Research Participant Assessment Score (RPA Comprehension) was a 17-item questionnaire designed to assess comprehension of study information at screening (Visit 6, week 12) between MICT and LASST trial designs. The same 17-item questionnaire was administered to the adolescent participant and to the caregiver participant. The items were scored as 1=incorrect, 2=partially correct, 3=correct (minimum possible score=17 and maximum possible score=51). Scores were assigned by two trained coders who independently listed to audio recordings of the RPA Comprehension questionnaire administration. Scores from the two coders were averaged for a final score. Higher scores indicate better comprehension. Mean (95% Confidence Interval) are the outcome measure reported.
Time Frame: Final Visit (Visit 6, Week12)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 53 | 25
Scores on a scale | 41.22 [39.88 to 42.55] | 41.27 [39.29 to 43.25]

4. Secondary Outcome: Caregiver Research Participant Assessment Score at Study End (Visit 6, Week 12)
Description: as for outcome 3
Time Frame: Final Visit (Visit 6, Week12)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 53 | 25
Scores on a scale | 43.28 [42.33 to 44.23] | 41.08 [39.67 to 42.49]

5. Secondary Outcome: Asthma Control Test Scores at Screening (Visit 1, Week -8)
Description: The Asthma Control Test is a 5-item Likert scale questionnaire; Scaling of items 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled); The score for each item is summed to generate a total score. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
  The study was powered to have greater than 90% power to detect a clinically meaningful difference of 3 in the ACT score between the MICT Trial Design and the LASST trial Design , assuming a mean score of 19 with a standard deviation of 4 (data from a previous ALA-ACRC trial).
Time Frame: Screening (Visit 1, week -8)
Population: The participant data set includes all participants who were randomized in each arm, the MICT trial design or LASST trial design. One participant in the MICT trial arm who was randomized to treatment at Visit 3 did not complete the study through Visit 6. The last available ACT score was used for this participant.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 54 | 25
scores on a scale | 22 [22 to 24] | 22 [21 to 23]

6. Secondary Outcome: Asthma Control Test Score at Final Visit (Visit 6, Week12)
Description: as for outcome 5
Time Frame: Final Visit (Visit 6, Week 12)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 54 | 25
scores on a scale | 24 [22 to 25] | 23 [22 to 24]

7. Secondary Outcome: Spirometry Quality Control Grade
Description: Spirometry grade scores in MICT participants (who performed spirometry at home) were compared with spirometry grade scores in LASST participants (who performed spirometry at the study sites). Spirometry grade scores were only available for LASST participants at Visit 3 (week 0), therefore only spirometry grade scores from Visit 3 were compared between MICT and LASST participants. Per the LASST trial no scoring was performed on the LASST participants for any other visit; the scoring for the LASST trial was for quality control only and was not a pre-specified trial outcome.
  Spirometry grade score scale was: 4.00 (highest=best possible score), 3.00, 2.00, 1.00, 0.00 (lowest=worst possible score). The maximum score was 4.00, the minimum score was 0.00. Higher scores indicate better spirometry score and therefore better quality.
Time Frame: Visit 3 (week 0)
Population: Twenty percent (20%) of available participant scores from Visit 3 (week 0) were randomly selected for analysis; N=11 participant scores were selected from the MICT Trial (20% of 54 scores =11). Eleven (11) participant scores were randomly selected from the LASST trial for analysis.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 11 | 11
scores on a scale | 3.75 [3.75 to 4.00] | 4.00 [4.00 to 4.00]

8. Secondary Outcome: Number of Errors in Questionnaires Completed by Participants at Visit 1 (Week -8).
Description: This outcome was to measure differences in timeliness and completeness of forms completed at home through REDCap in MICT participants compared with LASST participants.
  No data were collected for this outcome. This is because in designing the REDCap database used to send questionnaires to the MICT trial participants and to store the responses from the completed questionnaires, data checks were put into place to prevent incomplete forms. We did this by requiring all fields to be completed before the questionnaire could be submitted. If a questionnaire was not submitted, the study coordinator re-sent the questionnaire to the participant and the questionnaire was completed during the FaceTime visit. For the LASST participants, the study coordinator reviewed all forms the participant completed at the study site visit and any incomplete fields were completed at the time of the study site visit.
Time Frame: Visit 1 (week -8)
Population: No data were collected for this outcome.
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Errors in Questionnaires Completed by Participants at Visit 2 (Week -4).
Description: as for outcome 8
Time Frame: Visit 2 (week -4)
Population: No data were collected for this outcome.
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Errors in Questionnaires Completed by Participants at Visit 3 (Week 0).
Description: as for outcome 8
Time Frame: Visit 3 (week 0)
Population: No data were collected for this outcome.
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Errors in Questionnaires Completed by Participants at Visit 4 (Week 3).
Description: as for outcome 8
Time Frame: Visit 4 (week 3)
Population: No data were collected for this outcome.
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Errors in Questionnaires Completed by Participants at Visit 5 (Week 6).
Description: as for outcome 8
Time Frame: Visit 5 (week 6)
Population: No data were collected for this outcome.
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Errors in Questionnaires Completed by Participants at Visit 6 (Week 12).
Description: as for outcome 8
Time Frame: Visit 6 (week 12)
Population: No data were collected for this outcome.
Arm/Group | MICT Trial Design | LASST Trial Design
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were recorded starting the visit after treatment randomization at Visit 3 to Visit 6 for a period of 12 weeks in both the MICT and LASST trial.
Description: The data form used to collect adverse events specified specific symptoms that were most likely thought to occur in patients with asthma. In addition, the form listed specific new diagnoses that were thought most likely to occur in the study population. Lastly, the form included 4 fields to list any new symptom or diagnosis that was not previously specified on the form. If a subject experienced more than 1 of a given AE, the subject is counted only once for that AE.
Arm/Group | MICT Trial Design | LASST Trial Design
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/53 | 1/25
Other Adverse Events (participants affected / at risk) | 42/53 | 10/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MICT Trial Design (N=53) | LASST Trial Design (N=25)
acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Participant was scheduled for planned cholecystectomy and while hospitalized had significant post operative pain and developed acute chest syndrome.
Unsteady gait (Nervous system disorders) | 1 (1) | 0 (0) — Patient complained of headache lasting several weeks then developed unsteady gait. Hospitalized and given IV fluids, Toradol and Compazine with complete resolution at discharge.
Suicidality (Psychiatric disorders) | 0 (0) | 1 (1) — Participant expressed hopelessness, despair, and thoughts of suicide to her guidance counselor. She was admitted to the hospital under the Baker Act for 72 hours. Followup with psychiatrist as an outpatient.
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MICT Trial Design (N=53) | LASST Trial Design (N=25)
Skin bruising (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 19 (29) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 1 (1)
Chest pain (Cardiac disorders) | 15 (24) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (48) | 3 (3)
Muscle or joint pain (Musculoskeletal and connective tissue disorders) | 9 (14) | 1 (1)
Headache (General disorders) | 22 (43) | 4 (4)
Increased or irregular heartbeat (Cardiac disorders) | 7 (8) | 0 (0)
Restlessness or nervousness (Nervous system disorders) | 6 (12) | 0 (0)
Tremor (Nervous system disorders) | 6 (12) | 0 (0)
Runny nose and congestion (Respiratory, thoracic and mediastinal disorders) | 24 (45) | 2 (2)
Nausea and/or vomiting (Gastrointestinal disorders) | 9 (10) | 1 (1)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Allocation to trial type was not randomized; enrollment in LASST began 1 year before MICT, and LASST enrollment was competitive across the network. Parents and adolescents likely had varying cognitive abilities and experience with e-learning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (8):
  • Study Protocol (2016-08-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT02061280/Prot_000.pdf
  • Statistical Analysis Plan (2011-10-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT02061280/SAP_001.pdf
  • Informed Consent Form: 12-17 Assent LASST (2015-09-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT02061280/ICF_002.pdf
  • Informed Consent Form: PPF LASST (2015-09-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT02061280/ICF_003.pdf
  • Informed Consent Form: 12-17 Assent LASST RPA Ancillary (2014-04-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT02061280/ICF_004.pdf
  • Informed Consent Form: ICF-PPF LASST RPA Ancillary (2014-04-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT02061280/ICF_005.pdf
  • Informed Consent Form: 12-17 Assent MICT (2016-02-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT02061280/ICF_006.pdf
  • Informed Consent Form: ICF-PPF_MICT (2016-02-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT02061280/ICF_007.pdf